CLINICAL TRIAL: NCT00297232
Title: An Open-Label, Multicenter, Extension Study to Evaluate the Safety and Tolerability of Natalizumab Following Re-Initiation of Dosing in Multiple Sclerosis Subjects Who Have Completed Study C-1801, C-1802, C-1803, or C-1808 and a Dosing Suspension Safety Evaluation
Brief Title: Natalizumab (Tysabri) Re-Initiation of Dosing
Acronym: STRATA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-MS-321
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2015-05

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Natalizumab (Experimental): 300 mg intravenous (IV) infusions once every 4 weeks for up to 480 weeks
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab
  Other Names: Tysabri (BG00002)

SUMMARY:
The primary objectives for the initial treatment period of this study are to further evaluate the safety of natalizumab monotherapy by evaluating the risk of hypersensitivity reactions and immunogenicity following re-exposure to natalizumab and confirming the safety of switching from interferon (IFN), glatiramer acetate, or other multiple sclerosis (MS) therapies to natalizumab. The primary objective for the long-term treatment period of this study is to evaluate the long-term impact of natalizumab monotherapy on the progression of disability measured by Expanded Disability Status Scale (EDSS) changes over time.

DETAILED DESCRIPTION:
Study 101-MS-322 (NCT00306592) was conducted to evaluate the safety of natalizumab monotherapy following re-exposure to natalizumab in former clinical trial participants in Studies C-1801 (NCT00027300), C-1802 (NCT00030966), and C-1803 (NCT00097760) and included subjects in North America. In parallel with the conduct of that study, this study (101-MS-321 [NCT00297232]) was initiated for participants in Europe and the rest of the world. In addition, after 48 weeks, participants from 101-MS-322 (NCT00306592) could enter study 101-MS-321 (NCT 00297232), which was considered the Long-Term Treatment Period of 101-MS-322 (NCT00306592).

The primary purpose and primary outcome for both studies are identical; therefore, the combined long-term data from both studies are presented. (Combined Week 48 data from both studies are presented in the 101-MS-322 [NCT00306592] record.)

ELIGIBILITY:
Key Inclusion Criteria

* MS subjects who completed Study C-1801 (NCT00027300), C-1802 (NCT00030966), or C-1803 (NCT00097760) and a Dosing Suspension Safety Evaluation (neurological examination or a magnetic resonance imaging scan) or participated in the IMA 04001 (STARS) Study
* Subjects who are considered by the Investigator to be free of signs and symptoms suggestive of progressive multifocal leukoencephalopathy and willing to discontinue and remain free from concomitant immunosuppressive or immunomodulatory treatment (including IFN-beta and glatiramer acetate) while being treated with natalizumab during the study.
* In addition, subjects who completed 48 weeks of treatment in Study 101-MS-322 (NCT00306592) in Canada will be allowed to enter this study at the start of the long-term treatment period (Week 52 - 480).

Key Exclusion Criteria

* Considered by the Investigator to be immunocompromised
* History of persistent anti-natalizumab antibodies, based upon testing from prior natalizumab studies
* History of any major disease or malignancy
* Discontinued natalizumab in a previous study due to allergic reaction

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1094 (Actual)
Dates: Start 2006-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (98):
- Australia (3):
  - Research Site, Camperdown
  - Research Site, Heidelberg
  - Research Site, Parkville
- Belgium (6):
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Diepenbeek
  - Research Site, Melsbroek
  - Research Site, Sijsele
- Canada (10):
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, New York, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- Czechia (7):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Pardubice
  - Research Site, Pilsen
  - Research Site, Prague
- Denmark (3):
  - Research Site, Aarhus C
  - Research Site, Copenhagen
  - Research Site, Esbjerg
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Tampere
  - Research Site, Turku
- France (13):
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Clermont-Ferrand
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Nancy
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (10):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Giessen
  - Research Site, Hanover
  - Research Site, Hennigsdorf
  - Research Site, München
  - Research Site, Offenbach
  - Research Site, Osnabrück
  - Research Site, Regensburg
  - Research Site, Rostock
- Research Site, Athens, Greece
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Nyíregyháza
  - Research Site, Székesfehérvár
- Research Site, Dublin, Ireland
- Israel (2):
  - Research Site, Jerusalem
  - Research Site, Tel Litwinsky
- Italy (4):
  - Research Site, Bari
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Roma
- Netherlands (6):
  - Research Site, 's-Hertogenbosch
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Nieuwegein
  - Research Site, Nijmegen
  - Research Site, Rotterdam
- New Zealand (2):
  - Research Site, Auckland
  - Research Site, Christchurch
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Warsaw
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Málaga
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Stockholm
- Research Site, Basel, Switzerland
- Turkey (Türkiye) (2):
  - Research Site, Ankara
  - Research Site, Istanbul
- United Kingdom (7):
  - Research Site, Essex
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Newcastle upon Tyne
  - Research Site, Oxford
  - Research Site, Sheffield
  - Research Site, Stoke-on-Trent

REFERENCES:
- [Result] Gorelik L, Lerner M, Bixler S, Crossman M, Schlain B, Simon K, Pace A, Cheung A, Chen LL, Berman M, Zein F, Wilson E, Yednock T, Sandrock A, Goelz SE, Subramanyam M. Anti-JC virus antibodies: implications for PML risk stratification. Ann Neurol. 2010 Sep;68(3):295-303. doi: 10.1002/ana.22128. PMID 20737510
- [Result] Rudick RA, O'Connor PW, Polman CH, Goodman AD, Ray SS, Griffith NM, Jurgensen SA, Gorelik L, Forrestal F, Sandrock AW, Goelz SE. Assessment of JC virus DNA in blood and urine from natalizumab-treated patients. Ann Neurol. 2010 Sep;68(3):304-10. doi: 10.1002/ana.22107. PMID 20737514
- [Result] O'Connor P, Goodman A, Kappos L, Lublin F, Polman C, Rudick RA, Hauswirth K, Cristiano LM, Forrestal F, Duda P. Long-term safety and effectiveness of natalizumab redosing and treatment in the STRATA MS Study. Neurology. 2014 Jul 1;83(1):78-86. doi: 10.1212/WNL.0000000000000541. Epub 2014 Jun 4. PMID 24898925
- See also: The website of the National Multiple Sclerosis Society, an organization dedicated to providing information to individuals with MS, their families, and healthcare providers. — http://www.nationalmssociety.org
- See also: MSActiveSource.com is a resource for news, information, and disease management for all individuals touched by multiple sclerosis. This site is sponsored by Biogen Idec. — http://www.msactivesource.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants from studies 101-MS-321 (NCT00297232) and 101-MS-322 (NCT00306592) are included in this presentation of combined final data.
  Note: In the Participant Flow table, 'progressive multifocal leukoencephalopathy' is abbreviated to 'PML'. and John Cunningham virus is abbreviated to 'JCV'.
Period: Overall Study
Arm/Group | Natalizumab
Started | 1094
Completed | 489
Not Completed | 605
Not completed — Lack of Efficacy | 7
Not completed — Lost to Follow-up | 10
Not completed — Adverse Event | 63
Not completed — Voluntary Withdrawal | 120
Not completed — Subject was Noncompliant | 9
Not completed — Death | 9
Not completed — Anti-natalizumab Positive | 8
Not completed — Switched to Commercial Tysabri | 22
Not completed — Disease Progression | 8
Not completed — Fear of PML | 10
Not completed — Anti-JCV Antibody Positive | 13
Not completed — Miscellaneous | 5
Not completed — Sponsor Decision | 34
Not completed — Subject Relocated | 7
Not completed — Subject Withdrew Consent | 37
Not completed — Persistently Positive Antibodies | 11
Not completed — Investigator Withdrew From Program | 19
Not completed — Did Not Enroll to Week 264 | 34
Not completed — Did Not Enroll to Week 480 | 17
Not completed — No data available after Week 264 | 161
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Groups:
- Natalizumab: 300 mg IV infusions once every 4 weeks for up to 480 weeks
Arm/Group | Natalizumab
Number analyzed (Participants) | 1094
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (8.12)
Age, Customized [Number; unit: years]
  20 to 29 years | 98
  30 to 39 years | 347
  40 to 49 years | 454
  50 to 59 years | 195
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 755
  Male | 339

OUTCOME MEASURES:

1. Primary Outcome: Time to 24-week Confirmed Expanded Disability Status Scale (EDSS) Progression
Description: Time to 24-week confirmed EDSS progression in participants with at least 2 post-baseline milestone EDSS assessments. EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was reported. Confirmed 24-week EDSS progression was defined as ≥ 0.5 point increase from a baseline EDSS ≥ 6.0, or ≥ 1.0 point increase from a baseline EDSS ≥ 1.0 and < 6.0, or ≥ 1.5 point increase from a baseline EDSS of 0, all sustained for 24 weeks.
Time Frame: up to 480 weeks
Population: Participants with EDSS progression (regardless of length of follow-up) sustained for 24 weeks.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Natalizumab
Number analyzed (Participants) | 220
weeks | 121.9 [67.9 to 216.1]

2. Primary Outcome: Time to 48-week Confirmed EDSS Progression
Description: Time to 48-week confirmed EDSS progression in particpants with at least 2 post-baseline milestone EDSS assessments. EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was reported. Confirmed 48-week EDSS progression was defined as ≥ 0.5 point increase from a baseline EDSS ≥ 6.0, or ≥ 1.0 point increase from a baseline EDSS ≥ 1.0 and < 6.0, or ≥ 1.5 point increase from a baseline EDSS of 0, all sustained for 48 weeks.
Time Frame: up to 480 weeks
Population: Participants with EDSS progression (regardless of length of follow-up) sustained for 48 weeks.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Natalizumab
Number analyzed (Participants) | 181
weeks | 130.1 [72.4 to 216.1]

3. Primary Outcome: Time to 24-week Confirmed EDSS Improvement Where Baseline ≥ 2.0
Description: Time to 24-week confirmed EDSS improvement in subjects with at least 2 post-baseline milestone EDSS assessments. EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was reported. Confirmed 24-week EDSS improvement is defined as ≥ 1.0 point decrease from baseline sustained for 24 weeks.
Time Frame: Up to 480 weeks
Population: Participants with EDSS improvement (regardless of length of follow-up) sustained for 24 weeks.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Natalizumab
Number analyzed (Participants) | 173
weeks | 48.1 [24.1 to 119.9]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were collected from screening through the follow-up (492 weeks). Non-serious AEs were collected from baseline through Week 264.
Arm/Group | Natalizumab
Serious Adverse Events (participants affected / at risk) | 231/1094
Other Adverse Events (participants affected / at risk) | 752/1094
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab (N=1094)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 18
Urinary tract infection (Infections and infestations) | 13
Pneumonia (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 3
Bronchitis viral (Infections and infestations) | 2
Cystitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Epididymitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Hepatitis A (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Lower respiratory tract infection viral (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Meningitis viral (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pelvic inflammatory disease (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pneumonia streptococcal (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adenocarcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebellopontine angle tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Coombs negative haemolytic anaemia (Blood and lymphatic system disorders) | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 1
Immune reconstitution inflammatory syndrome (Immune system disorders) | 11
Anaphylactic shock (Immune system disorders) | 2
Hypersensitivity (Immune system disorders) | 2
Anaphylactic reaction (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Goitre (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 4
Suicide attempt (Psychiatric disorders) | 3
Completed suicide (Psychiatric disorders) | 2
Mania (Psychiatric disorders) | 2
Suicidal ideation (Psychiatric disorders) | 2
Abnormal behaviour (Psychiatric disorders) | 1
Anxiety disorder (Psychiatric disorders) | 1
Bipolar I disorder (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 21
Multiple sclerosis (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 2
Trigeminal neuralgia (Nervous system disorders) | 2
Altered state of consciousness (Nervous system disorders) | 1
Amnesia (Nervous system disorders) | 1
Cerebral cyst (Nervous system disorders) | 1
Cerebrovascular insufficiency (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Facial neuralgia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Eye swelling (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Retinal tear (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Myocardial fibrosis (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Peripheral ischaemia (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Venous stenosis (Vascular disorders) | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 3
Abdominal adhesions (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Anal fissure (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 2
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Rectal prolapse (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 5
Cholecystitis (Hepatobiliary disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Melanocytic hyperplasia (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Renal colic (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 1
Neurogenic bladder (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1
Metrorrhagia (Reproductive system and breast disorders) | 2
Uterine polyp (Reproductive system and breast disorders) | 2
Adnexal torsion (Reproductive system and breast disorders) | 1
Breast hyperplasia (Reproductive system and breast disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Rectocele (Reproductive system and breast disorders) | 1
Vaginal prolapse (Reproductive system and breast disorders) | 1
Congenital anomaly (Congenital, familial and genetic disorders) | 1
Pyrexia (General disorders) | 2
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Multi-organ failure (General disorders) | 1
Oedema (General disorders) | 1
Pain (General disorders) | 1
Polyp (General disorders) | 1
Blood pressure increased (Investigations) | 1
Polyomavirus test positive (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 7
Head injury (Injury, poisoning and procedural complications) | 4
Lower limb fracture (Injury, poisoning and procedural complications) | 3
Concussion (Injury, poisoning and procedural complications) | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2
Road traffic accident (Injury, poisoning and procedural complications) | 2
Wrist fracture (Injury, poisoning and procedural complications) | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Face injury (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Gun shot wound (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Peripheral nerve decompression (Surgical and medical procedures) | 1
Spinal laminectomy (Surgical and medical procedures) | 1
Thyroid nodule removal (Surgical and medical procedures) | 1
Vascular graft (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab (N=1094)
Diarrhoea (Gastrointestinal disorders) | 80
Fatigue (General disorders) | 102
Nasopharyngitis (Infections and infestations) | 256
Upper respiratory tract infection (Infections and infestations) | 192
Urinary tract infection (Infections and infestations) | 162
Influenza (Infections and infestations) | 122
Sinusitis (Infections and infestations) | 82
Bronchitis (Infections and infestations) | 67
Fall (Injury, poisoning and procedural complications) | 61
Back pain (Musculoskeletal and connective tissue disorders) | 113
Arthralgia (Musculoskeletal and connective tissue disorders) | 86
Pain in extremity (Musculoskeletal and connective tissue disorders) | 62
Multiple sclerosis relapse (Nervous system disorders) | 164
Headache (Nervous system disorders) | 157
Dizziness (Nervous system disorders) | 62
Depression (Psychiatric disorders) | 72

LIMITATIONS AND CAVEATS:
Sponsor decided to terminate the study prior to all subjects reaching Week 480 as the primary objective was deemed to have been met and only approximately 45% of the original STRATA population remained in the study at the time of study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.